CLINICAL TRIAL: NCT00730249
Title: Quality Assurance of Administering Methylphenidate in Adults With ADHD
Brief Title: Quality Assurance of Administering Methylphenidate in Adults With Attention Deficit Hyperactivity Disorder (ADHD) - QUMEA
Acronym: QUMEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medice Arzneimittel Pütter GmbH & Co KG (Industry)
Responsible Party: Dr. Roland Fischer/Head of Medical Dept., Medice Arzneimittel Pütter GmbH & Co. KG
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6520-0650-13
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Attention Deficit Hyperactivity Disorder; adult; methylphenidate hydrochloride; Medikinet retard; controlled clinical trial; safety; randomized, double-blind, placebo-controlled trial; treatment; central nervous system stimulants; therapeutic uses
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: methylphenidate hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: methylphenidate hydrochloride — sustained release, twice daily, dosage according to an individual titration schedule
  Other Names: Medikinet retard
  Arms: 1
Drug: Placebo — twice daily according to an individual titration schedule
  Arms: 2

SUMMARY:
Investigation of efficacy of high-dose extended-release Methylphenidate in adults with ADHD, compared with a placebo

ELIGIBILITY:
Inclusion Criteria:

* patient treated as out-patient
* score of 85 or greater in IQ-test (MWT-B)
* diagnosis of ADHD according ADHS-CL (DSM IV) and WRAADDS > 35 points
* ADHD symptoms have existed since childhood (WURS-k >= 30)
* Body Mass Index >= 20 and body weight < 130 kg
* willing to eat breakfast and lunch
* patient is willing and able to come to the observation appointments
* written consent of the patient to participate in the study

Exclusion Criteria:

* treatment with psychostimulants in the past two weeks before screening
* shift work or night work
* alcohol, medication or drug dependency in the past six months or manifest drug abuse
* diagnosis of a psychosis (SKID-I)
* epileptic attacks in the past
* EEG result which suggests epilepsy
* acute depressive episode according to ICD-10 F32.2 and ICD-10 F32.3 (Beck-Depression-Inventory > 18)
* Illness with schizophrenic symptoms (SKID-I)
* acute manic episode, bipolar disorder(SKID-I)
* diagnosis of a tic disorder
* acute anorexia
* acute prominent panic disorder and generalised anxiety (SKID-I)
* clinically relevant kidney disorders
* creatinine > 1,5 x upper norm-range
* clinically relevant liver disorder
* SGOT and/or SGPT > 2 x upper norm-range
* pathological ECG-finding
* QTc > 450 msec in male, QTc > 470 msec in female
* high blood pressure (anamnesis or blood pressure > 140/90 mm Hg at screening)
* known acclusive arterial disease
* angina pectoris (anamnesis or ECG-finding)
* cardiac arrhythmias (anamnesis or ECG-finding)
* KHK (anamnesis or ECG-finding)
* post heart-attack status (anamnesis or ECG-finding)
* post stroke status
* known elevated intra-ocular pressure
* known enlarged prostates
* latent and manifest hyperthyreosis
* TSH < lower norm-range
* patient with a terminal disease (e.g. cancer)
* participation in a clinical study within the past 30 days
* participation in this study at an earlier point in time
* simultaneous participation in another clinical trial
* women of child-bearing age without adequate contraception (contraceptives, intrauterine device , no sexual intercourse)
* pregnancy (positive pregnancy test) or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Wender-Reimherr Adult Attention Deficit Disorder Scale (WRAADDS) in last study-week (Placebo vs. Verum, double-blind phase, week 6) | 20 weeks

SECONDARY OUTCOMES:
CAARS-Self-Report: Long Version (CAARS-S:L) | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland Fischer, Dr., Study Chair — Medice Arzneimittel Pütter GmbH & Co KG; Michael Rösler, Prof. Dr., Study Director — Universität des Saarlandes, Institut für gerichtliche Psychiatrie
Locations (11):
- Germany (11):
  - Praxis Johannes Fuhr, Bad Wildungen
  - Charité Campus Mitte, Station 155, Berlin
  - Gemeinschaftspraxis für Kinder- und Jugendpsychiatrie, Psychotherapie, Berlin
  - Universitätsklinik Bochum, Bochum
  - Universitätsklinikum Freiburg, Abteilung für Psychiatrie und Psychotherapie, Freiburg im Breisgau
  - Universitäts-Klinik Eppendorf,, Hamburg
  - Praxis Dr. Heinrich Goossens-Merkt, Hamburg
  - Universität des Saarlandes, Institut für gerichtliche Psychiatrie, Homburg
  - Praxis Thomas Wirth, Ludwigsburg
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Medizinisches Studienzentrum Würzburg, Würzburg